CLINICAL TRIAL: NCT01728896
Title: A Randomized Controlled Trial of Patient-Initiated and ConTrolled Oral Refeeding in Acute Pancreatitis
Brief Title: Patient-Initiated and ConTrolled Oral Refeeding (PICTOR)
Acronym: PICTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Max Petrov, Prinicpal Investigator Dr. Max Petrov, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: NTX/12/06/051
Record Dates: First submitted 2012-11-05; First posted 2012-11-20 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Acute Pancreatitis
Keywords: Acute pancreatitis, nutrition
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient-controlled oral refeeding (Experimental): Patients will be allowed to drink and eat hospital food freely as tolerated.
  Interventions: Other: Patient-controlled oral refeeding
- Conventional management (No Intervention)

INTERVENTIONS:
Other: Patient-controlled oral refeeding
  Arms: Patient-controlled oral refeeding

SUMMARY:
The first step in treating patients with acute pancreatitis is to provide pain relief and intravenous fluids to keep them comfortable. As the pain subsides and patient starts to feel better food and fluids by mouth are restarted. This is done to rest the pancreas which is the organ that has been inflamed.

In some patients when food by mouth restarts they have pain and as a consequence they have a longer stay in hospital. It is thought that patients who have little pain and are within 24 hours of admission to hospital do well if they control their own food intake. This is in contrast to the usual treatment where the treating team advise when eating should restart.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of acute pancreatitis
* age > 18 years
* written informed consent

Exclusion Criteria:

* ongoing need for opiates
* >96 hours after onset of symptoms
* chronic pancreatitis
* post-ERCP pancreatitis
* intraoperative diagnosis
* pregnancy
* malignancy
* received nutrition before randomisation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Oral food intolerance | Participants will be followed for the duration of hospital stay, an expected average of 7 days

SECONDARY OUTCOMES:
Time from admission until tolerance of oral food | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Total length of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Need for opiates | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Need for opiates is defined when one (or more) of the following has been administered:
  * Codeine phosphate
  * Fentanyl
  * Morphine, Sevredol, Meslon
  * Oxynorm, Oxycodone
  * Tramadol
Change in pain intensity | Baseline and 24, 48, 72h after randomisation
Progression of acute pancreatitis severity | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  To be defined according to the 2012 determinant-based classification of acute pancreatitis severity
Hospital readmission | 2 weeks after hospital discharge
Local and systemic complications | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  To be defined according to the 2012 determinant-based classification of acute pancreatitis severity
Number and type of interventions during hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Time from admission until first flatus | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Change in blood glucose | Baseline and 24, 48, 72h after randomisation
Change in plasma C-reactive protein | Baseline and 24, 48, 72h after randomisation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Auckland; Auckland City Hospital, Auckland, New Zealand